CLINICAL TRIAL: NCT03420313
Title: Interim Buprenorphine Treatment to Bridge Waitlist Delays: Stage II Evaluation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Stacey C. Sigmon, Associate Professor, UVM Dept of Psychiatry, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA042790-01 (NIH)
Record Dates: First submitted 2017-12-19; First posted 2018-02-05 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Opioid-use Disorder
Keywords: buprenorphine; waitlist; interim treatment; opioid use disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Intervention Model Description: randomized parallel two-group trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interim Buprenorphine Treatment (Experimental): Interim Buprenorphine Treatment includes (a) Maintenance treatment with Buprenorphine/ naloxone sublingual tablets with bi-monthly clinic visits for observed dosing and the remaining doses dispensed at home via a secure computerized portable device (Med-O-Wheel, Addoz, Finland).
  (b) nightly calls from an automated Interactive Voice Response (IVR) phone system to assess any drug use, withdrawal and craving, (c) IVR-generated random call-backs for urinalysis and pill counts, and (d) HIV+Hepatitis education delivered via iPad. (e) monthly follow-up assessments
  Interventions: Drug: Buprenorphine/naloxone sublingual tablets
- Waitlist Control (No Intervention): Waitlist Control participants will remain on the waitlist for their treatment of choice but complete the same monthly assessments.

INTERVENTIONS:
Drug: Buprenorphine/naloxone sublingual tablets — 24-week maintenance with buprenorphine/naloxone sublingual tablets (plus other technology-assisted components described previously)
  Other Names: BUP
  Arms: Interim Buprenorphine Treatment

SUMMARY:
Despite the demonstrated effectiveness of agonist treatment for opioid dependence and alarming recent increases in overdose deaths, waiting lists for treatment persist. In a Behavioral & Integrative Treatment Development pilot study, the investigators demonstrated the initial efficacy a novel Interim Buprenorphine Treatment (IBT) to mitigate the risks (e.g., illicit opioid use, IV drug use) associated with treatment delays. However, consistent with that R34 mechanism, our initial pilot study involved a limited sample size and was conducted at a single academic, well-controlled research clinic with an extensive history of research. It is important to replicate these very positive pilot results and begin to evaluate whether they generalize to less-controlled rural environments that are being so adversely impacted by the current opioid abuse epidemic. In this Stage II randomized parallel two-group trial, the investigators will evaluate the efficacy of IBT using a larger sample of 100 waitlisted opioid-dependent adults (50 IBT, 50 WLC). UVM will serve as the coordinating center and we will aim to partner with health centers and other convenience sites in rural Vermont counties to conduct study visits while overcoming barriers commonly encountered in rural areas (e.g., transportation issues, socioeconomic barriers). The proposed research builds directly on the promising Stage I results and has the potential to substantially reduce the vast individual and societal costs associated with opioid treatment delays.

DETAILED DESCRIPTION:
Despite the demonstrated effectiveness of agonist treatment for opioid dependence and alarming recent increases in overdose deaths, waiting lists for treatment persist. Opioid-dependent individuals can remain on waitlists for months, during which they are at substantial risk for illicit drug use, criminal activity, infectious disease, overdose and premature death. One effort to reduce these risks has been to extend interim methadone treatment (IMT; i.e., daily methadone without counseling) to individuals awaiting entry into a methadone program. IMT significantly reduces illicit opioid use and criminality during treatment delays. However, it is limited to licensed specialty clinics, requires daily visits, prohibits take-home doses and cannot exceed a 120-day duration. These regulatory restrictions have constrained the widespread use of IMT.

With a Behavioral & Integrative Treatment Development R34, the investigators have developed a novel Interim Buprenorphine Treatment (IBT) to mitigate the risks associated with treatment delays while surmounting the limitations noted above for methadone. It includes key components to permit delivery of potentially life-saving pharmacotherapy while minimizing nonadherence: (a) Buprenorphine (BUP) offers a regulatory and safety profile that is uniquely compatible with interim dosing. Participants receive BUP maintenance with bi-monthly clinic visits and the remaining doses dispensed at home via a secure computerized portable device (Med-O-Wheel, Addoz, Finland). Participants also receive (b) nightly calls from an automated Interactive Voice Response (IVR) phone system to assess any drug use, withdrawal and craving, (c) IVR-generated random call-backs for urinalysis and pill counts, and (d) HIV+Hepatitis education delivered via iPad.

Our Stage I pilot data strongly support the initial efficacy of this intervention. Among 50 waitlisted opioid-dependent adults randomized to IBT (n=25) or Waitlist Control (WLC; n=25) conditions for 12 weeks, 85%, 84% and 68% of IBT participants are abstinent at 4, 8 and 12-week assessments vs. 0%, 0% and 0% of WLC participants (p<.001). IBT participants also reported significantly greater reductions in illicit opioid use and IV drug use frequency and completing 96% of daily IVR calls and random call-backs. These outcomes represented a substantial first step towards the development of an intervention that can reduce individual and societal risks during delays to conventional treatment.

However, consistent with the R34 mechanism, our initial pilot study involved a limited sample size and was conducted at a single academic, well-controlled research clinic with an extensive history of research and a brief treatment duration. It is important to replicate these very positive pilot results and begin to evaluate whether they generalize to less-controlled rural environments that are being so adversely impacted by the current opioid abuse epidemic as well as over longer treatment durations. Important to underscore is that our IBT components (i.e., Med-O-Wheel, IVR, HIV+Hepatitis application) are highly transportable, which increases the potential of extending them to sites outside of the university setting while retaining efficacy.

Primary Aim: In this Stage II randomized parallel two-group trial, the investigators will evaluate the efficacy of IBT using a larger sample of 100 waitlisted opioid-dependent adults (50 IBT, 50 WLC). UVM will serve as the coordinating center and we will aim to partner with health centers and other convenience sites in rural Vermont counties to conduct study visits while overcoming barriers commonly encountered in rural areas (e.g., transportation issues, socioeconomic barriers). Participants randomized to IBT will receive the intervention described above for a duration of 24-weeks; WLC participants will remain on the waitlist for their treatment of choice but complete monthly assessments. It is hypothesized that IBT participants will achieve significantly greater illicit opioid abstinence relative to WLC participants.

The proposed research builds directly on the promising Stage I results and has the potential to substantially reduce the vast individual and societal costs associated with opioid treatment delays. By facilitating the eradication of waitlists, this project represents a significant departure from the status quo and stands to produce a fundamental shift in how treatment for opioid dependence is conceptualized and delivered.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion, participants must be >=18 years old, in good health, meet DSM-V criteria for opioid use disorder, provide an opioid-positive urine and be currently waitlisted with a community opioid treatment clinic or provider.

Exclusion Criteria:

* Those with a significant psychiatric or medical illness that may interfere with consent or participation will be excluded, as will those who are pregnant or nursing. Those dependent on sedative-hypnotics will be excluded, due to the medical risks and notably low success rates with sedative-dependent opioid abusers (Stitzer & Chutuape, 1999).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Illicit opioid abstinence | 12 weeks
  Overall percentage of urinalyses biochemically verified to be abstinent for illicit opioids during the treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sigmon SC, Peck KR, Batchelder SR, Badger GJ, Heil SH, Higgins ST. Technology-Assisted Buprenorphine Treatment in Rural and Nonrural Settings: Two Randomized Clinical Trials. JAMA Netw Open. 2023 Sep 5;6(9):e2331910. doi: 10.1001/jamanetworkopen.2023.31910. PMID 37755833